CLINICAL TRIAL: NCT05631028
Title: Effect of Dexmedetomidine Pretreatment on The Effective Dose of Remimazolam Tosilate Inhibiting Cardiovascular Response to Intubation of Double-Lumen Endobronchial Tubes: A Clinical Research
Brief Title: 95% Effective Dose(ED95) of Remimazolam During Dexmedetomidine Pretreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyou Wei (Other)
Responsible Party: Sponsor-Investigator, Shiyou Wei, Medical Master, Attending Doctor., Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2022LY0416
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Anesthesia Induction
Keywords: Anaesthetic; Remimazolam; Cardiovascular Reaction
MeSH Terms: conditions — Lung Neoplasms | interventions — Dexmedetomidine; Injections; Powders

STUDY DESIGN:
Intervention Model Description: This study is a clinical trial of dynamic design dose exploration evaluating the effect of dexmedetomidine pretreatment on the effective dose of remimazolam tosilate inhibiting cardiovascular response to intubation of double-lumen endobronchial tubes. Following the design principle, conduct dynamic exploration by sequential method, using the near ED95 drug dose for subjects according to the pretest.To determine whether the next subject increases or decreases the pre-set fixed drug dose according to the previous subject. The trial was stopped when seven exchange points occurred, at which point the total sample size was obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Dexmedetomidine pretreatment dose was 0. The effective dose of remimazolam tosilate inhibiting cardiovascular response during double-lumen tracheal intubation in elderly patients (age > 65 years) and young patients (18 < age <65 years) was explored respectively, without the use of dexmedetomidine. The starting dose of Remimazolam tosilate for Injection (36mg per bottle, powder, HengRui medicine, China) was 0.25 mg / kg, and the adjusted unit dose was 0.01mg.
  Interventions: Drug: Remimazolam tosilate
- Group B (Experimental): Dexmedetomidine hydrochloride injection (200ug per bottle, HengRui medicine, China) was diluted to 50ml and the pretreatment dose was 0.5μg/kg at first 10 mins.The starting dose of Remimazolam tosilate for Injection (36mg per bottle, powder, HengRui medicine, China) was 0.15 mg / kg, and the adjusted unit dose was 0.01mg.
  Interventions: Drug: Dexmedetomidine; Drug: Remimazolam tosilate
- Group C (Experimental): Dexmedetomidine hydrochloride injection (200ug per bottle, HengRui medicine, China) was diluted to 50ml and the pretreatment dose was 1μg/kg at first 10 mins.The starting dose of Remimazolam tosilate for Injection (36mg per bottle, powder, HengRui medicine, China) was 0.1 mg / kg, and the adjusted unit dose was 0.01mg.
  Interventions: Drug: Dexmedetomidine; Drug: Remimazolam tosilate

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is the most popular adjuvant to anesthesia. Groups was grouped according to different preadministered doses of dexmedetomidine. This allows a more comprehensive assessment of remimazolam under different use. Three groups were set separately, and Group A, Group B, and Group C correspond to 0,0.5, and 1 μg/kg at first 10 mins , respectively.
  Other Names: Dexmedetomidine hydrochloride injection (200ug per bottle, HengRui medicine, China)
  Arms: Group B; Group C
Drug: Remimazolam tosilate — Remimazolam tosilate has a short clinical time and a lack of combination with dexmedetomidine for dual-lumen endotracheal intubation. The optimal use dose of Remimazolam tosilate was explored separately from different dexmedetomidine doses.
  Other Names: Remimazolam tosilate for Injection (36mg per bottle, powder, HengRui medicine, China)

SUMMARY:
General anesthesia with double-lumen endobronchial tubes intubation is the main anesthesia method in thoracic surgery.However, double-lumen endobronchial tubes intubation can produce greater stimulation and cause more cardiovascular reactions, and the ideal anesthetic drugs can effectively reduce adverse reactions.Remimazolam is a new type of benzodiazepine drug that can be safely used for the induction and maintenance of general anesthesia, and it is an ideal and short-acting anesthetic alternative.As the new drug has had a short clinical entry time.There are few clinical data in all aspects, so it is necessary to clarify its rational use in the induction of anesthesia.Dexmedetomidine is a highly selective α 2 adrenergic receptor agonist, and it is currently the most popular adjunct to clinical anesthesia.However, the clinical data of anesthesia induction by dexmedetomidine combined with Remimazolam are rarely reported.

In the case of prior use of dexmedetomidine, to explore 50% effective dose (ED50) and ED95 of Remimazolam for the induction of anesthesia to inhibit the cardiovascular response of double-lumen bronchial intubation, in order to provide more data for the rational use of remimazolam and a reference for clinical rational drug use.

DETAILED DESCRIPTION:
This study is a clinical trial of adaptive design dose exploration evaluating the effect of dexmedetomidine pretreatment on the effective dose of remimazolam tosilate inhibiting cardiovascular response to intubation of double-lumen endobronchial tubes.Following the design principle, conduct dynamic exploration by sequential method, using the near ED95 drug dose for subjects according to the pretest.To determine whether the next subject increases or decreases the pre-set fixed drug dose according to the previous subject. The trial was stopped when seven exchange points occurred, at which point the total sample size was obtained.

For more detailed measures, please follow us below.

ELIGIBILITY:
Inclusion Criteria:

* Optional Video-Assisted Thoracoscopic Surgery (VATS)
* More than 18 years old
* American Association of Anesthesiologists (ASA) grade I~III

Exclusion Criteria:

* Systolic pressure ≥160 mmHg or diastolic pressure ≥110 mmHg or heart rate ≥ 110 beats / min in the operating room when quietly
* Long-term use of analgesia or sedation drugs before surgery
* Pregnancy, lactation, pregnancy possibility and planned pregnancy
* Allergy history of the test drug
* Mental illness or an inability to communicate normally.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
ED50 and ED95 of remimazolam | Through study completion, an average of 3 month.
  Half of the effective doses (ED50) and 95% effective doses (ED95 ) of remimazolam to inhibit the cardiovascular response of double-lumen bronchial intubation during anesthesia induction after dexmedetomidine (DEX) pretreatment.
  Positive cardiovascular responses is determined when the highest hypertension or heart rate caused by bronchial intubation exceeds 15% of the baseline value. And the test will be ended with seven positive to negative transitions through sequential dose exploration. ED50 and ED 95 will be calculated by probit regression using the collected dose and cardiovascular response outcome data after study completion.

SECONDARY OUTCOMES:
Cardiovascular response within 3 min of intubation | The evaluation time included the start of endotracheal intubation until three minutes after completion.
  The criteria of positive cardiovascular response to double-lumen bronchial intubation are the amplitude of mean arterial blood pressure (MAP) or heart rate (HR) fluctuations was 15% greater than the base value within 3 min after intubation . Or the patient had a tachycardia (heart rate ≥ 120 per min) or blood pressure increased more than 180 mmHg.
Blood Pressure | Intraoperative (Four time points. Time 1: When calm in the operating room. Time 2: At the end of dexmedetomidine pumping. Time 3: End of the remimazolam infusion. Time 4:the start of endotracheal intubation until 3 min after completion)
  Blood pressure (systolic, diastolic, mean arterial pressure) were used to evaluate cardiovascular response. The measurements were made by Philips Patient Monitor (IntelliVue MX800).
Heart Rate | Intraoperative (Four time points. Time 1: When calm in the operating room. Time 2: At the end of dexmedetomidine pumping. Time 3: End of the remimazolam infusion. Time 4:the start of endotracheal intubation until 3 min after completion)
  Heart rate(HR) were used to evaluate cardiovascular response, which was measured by Philips Patient Monitor (IntelliVue MX800).
Success rate of sedation | Through study completion, an average of 3 month.
  Whether sedation failure occurs during the exploration of an effective dose, As assessed by modified observer's assessment of alert /sedation scale (MOAA / S), when MOAA / S ≤2 indicates loss of consciousness, implying successful sedation. The success rate of sedation for each group will be calculated only after study completion.
Incidence of Hypotension | Through study completion, an average of 3 month.
  Systolic blood pressure < 90 mmhg or mean arterial pressure(MAP) < 60mmhg throughout the induction of anesthesia. At the entire anesthesia induction process , we measured blood pressure by patient monitor to compare whether hypotension occurred, but the incidence of hypotension will be calculated only after study completion.
The incidence of reduced heart rate | Through study completion, an average of 3 month.
  Heart rate < 50 per min throughout the induction of anesthesia. At the entire anesthesia induction process , we measured heart rate by patient monitor to compare whether reduced heart rate occurred, but the incidence of reduced heart rate will be calculated only after study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyou Wei, MD, Principal Investigator — Tongji University
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei S, Liu X, Chang R, Chen X, Zheng T, Wang J, Liu H, Zhang F, Song J, Lv X. Effect of pre-use of Dexmedetomidine on the effective inhibitory dose of remimazolam tosilate on positive cardiovascular response in double-lumen endobronchial intubation: a clinical study. BMC Anesthesiol. 2023 Nov 23;23(1):382. doi: 10.1186/s12871-023-02305-8. PMID 37996787